CLINICAL TRIAL: NCT04560309
Title: Role of Glutamine as Myocardial Protector in Elective On-Pump Coronary Artery Bypass Graft Surgery With Low Ejection Fraction
Brief Title: Role of Glutamine as Myocardial Protector in Elective On-Pump CABG Surgery With Low EF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, I Made Adi Parmana, MD, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/466/KEP059/202; LB.02.01/VII/466/KEP059/202 (Other: National Cardiovascular Center Harapan Kita Indonesia)
Record Dates: First submitted 2020-09-07; First posted 2020-09-23 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Bypass; Cardiopulmonary Bypass; Coronary Artery Disease
Keywords: Glutamine; Myocardial protection; Coronary artery bypass grafting; Cardiopulmonary bypass; Low ejection fraction; Myocardial injury
MeSH Terms: conditions — Coronary Artery Disease | interventions — alanylglutamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine (Experimental): Intravenous L-alanyl-L-glutamine 0.5 mg/kgbw
  Interventions: Drug: L-alanyl-L-glutamine dipeptide
- Control (Placebo Comparator): Intravenous NaCl 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-alanyl-L-glutamine dipeptide — Intravenous infusion of 0.5 mg/kgbw L-alanyl-L-glutamine dipeptide diluted in normal saline to volume of 500 mL, started after induction of anesthesia for 24 hours.
  Other Names: Dipeptiven
  Arms: Glutamine
Drug: Placebo — Intravenous infusion of 500 mL normal saline, started after induction of anesthesia for 24 hours.
  Other Names: Normal saline
  Arms: Control

SUMMARY:
Coronary artery disease has the highest mortality rate worldwide and coronary artery bypass grafting (CABG) is the most common cardiac surgery performed in patients with coronary artery disease to revascularize the heart. Despite of improvement in operation techniques, cardioplegia, cardiopulmonary bypass (CPB), myocardial injury related to on-pump CABG is still prominent. In patient with low ejection fraction undergone on-pump CABG, myocardial injury is related to worse outcome and prognosis during peri-operative and post-operative period. On-pump CABG patients with low ejection fraction has increased (up to four times higher) post-operative in hospital mortality rate compared to patient with normal ejection fraction. Administration of intravenous glutamine had been documented in reducing myocardial damage during cardiac surgery and previous studies indicated that glutamine can protect against myocardial injury by various mechanism during ischemia and reperfusion. The purpose of this study to determine whether intravenous glutamine could prevent the decline of plasma glutamine level, reduce myocardial damage, improve hemodynamic profile, and reduce morbidity of on-pump CABG in patients with low ejection fraction.

DETAILED DESCRIPTION:
The study was a double-blind randomized controlled trial to assess the role of glutamine as a myocardial protection during coronary artery bypass grafting under cardiopulmonary bypass in patients with left ventricle ejection fraction of 31-50%. This study was approved by Institutional Review Board of National Cardiovascular Center Harapan Kita and informed consent was obtained before randomization for patient eligible for this study. Allocation of participant to the treatment group was done by block randomization by staff who was not involved in the study. The intervention drug was prepared by pharmacist who also was not involved in the study. Glutamine solution was supplied as L-alanyl-L-glutamine dipeptide (Dipeptiven, 200 mg/mL, Fresenius Kabi, Bad Homburg, Germany) and was prepared to contain 0.5gr/kgbw glutamine diluted in NaCl 0.9% to a final volume of 500 mL. Placebo was supplied as 500 ml of NaCl 0.9%, prepared in similar fashion and packaging as glutamine solution. Principal investigator, care provider, outcome assessor, and participant were blinded to the assigned group until after the end of the study.

Baseline participant characteristics were collected before the intervention included age, sex, body weight, body height, body mass index, and documented pre-operative left ventricle ejection fraction. Coronary artery bypass grafting and cardiopulmonary bypass was done in concordance to standard operating procedure in National Cardiovascular Center Harapan Kita, followed by transit time flow meter measurement to ensure quality of the graft. Modifying factor of the study, the investigators measured duration of surgery, duration of cardiopulmonary bypass, and duration of aortic cross clamp.

The primary outcome of the study was plasma troponin I level. The investigators anticipated plasma troponin I level difference of 20% with standard deviation of 0.04 ng/mL, and for statistical power of 80% and level of significance of 0.05, the required sample size was 24.5 participants per group. As anticipation for participant drop out, the investigators planned to recruit a total of 60 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary heart disease indicated for elective coronary artery bypass grafting under cardiopulmonary bypass
* Patients with left ventricle ejection fraction 31% -50% confirmed by echocardiography or radio nuclear study.
* Patients age ≥18 years
* Never had heart surgery before
* Agree to participate in the study and signed informed consent

Exclusion Criteria:

* Emergency coronary artery grafting bypass
* Having additional procedures other than coronary artery bypass grafting
* History of myocardial infarction with onset less than 3 months
* Patients with serum creatinine level more than 2 g/dL
* Patients with ALT/AST levels more than 1.5 times the upper limit of normal value
* Required to use intra-aortic balloon pump pre-operatively
* History of stroke with onset less than 3 months
* History of pre-operative atrial fibrillation
* History of heart conduction problem and/or using a pacemaker
* Patients with HIV
* Contraindications to pulmonary artery catheter insertion

Drop out Criteria

* Experiencing stroke after surgery
* Experiencing surgery related complication (haemorrhage) requiring re operation
* Requiring continuous veno-venous hemofiltration or haemodialysis after surgery
* Delayed sternal closure
* Aortic cross clamp duration more than 120 minutes and/or cardiopulmonary bypass time more than 180 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I Made Adi Parmana, Principal Investigator — National Cardiovascular Center Harapan Kita Indonesia
Locations (1):
- National Cardiovascular Center Harapan Kita Hospital Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data reported in this study will be made available on request after publication and ending 36 months following article publication. Researchers needs to state their aims of analyses and provide a methodologically sound proposal. Proposals should be directed to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication until 36 months following article publication
Access Criteria: Researchers needs to state their aims of analyses and provide a methodologically sound proposal. Proposals should be directed to the corresponding author.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on inclusion criteria. This study was carried out at National Cardiovascular Center Harapan Kita. Written informed consent was obtained from all eligible patients. This study was conducted from January to October 2021.
Pre-assignment Details: Sixty patients with a left ventricle EF of 31-50% who underwent on-pump CABG were included in this study and randomized to treatment. Two patients were dropped out in this study
Period: Overall Study
Arm/Group | Glutamine | Control
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1
Not completed — Meet drop out criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glutamine | Control | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.21 (7.29) | 61.31 (6.48) | 60.76 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.25 (2.53) | 26.47 (2.85) | 26.36 (2.67)
Pre-op Ejection Fraction [Median (Full Range); unit: percent] | 41.44 [31.00 to 50.00] | 44.00 [31.00 to 49.00] | 43.00 [31.00 to 50.00]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Troponin I at Baseline
Description: Plasma troponin I were measured using enzyme immunoassay (ELISA) in unit of ng/mL
Time Frame: Before induction to anesthesia
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
ng/mL | 0.42 [0.00 to 27.00] | 0.17 [0.00 to 1.98]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.993, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05

2. Primary Outcome: Plasma Troponin I at 5 Minute After Cardiopulmonary Bypass
Description: Plasma troponin I were measured using enzyme immunoassay (ELISA) in unit of ng/mL
Time Frame: 5 minute after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
ng/mL | 1.72 (0.98) | 1.68 (1.10)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.883, Unpaired T-Test — The threshold for statistical significance was p < 0.05

3. Primary Outcome: Plasma Troponin I at 6 Hour After Cardiopulmonary Bypass
Description: Plasma troponin I were measured using enzyme immunoassay (ELISA) in unit of ng/mL
Time Frame: 6 hour after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
ng/mL | 3.43 (1.51) | 4.41 (1.89)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.034, Unpaired T-Test — The threshold for statistical significance was p < 0.05

4. Primary Outcome: Plasma Troponin I at 24 Hour After Cardiopulmonary Bypass
Description: Plasma troponin I were measured using enzyme immunoassay (ELISA) in unit of ng/mL
Time Frame: 24 hour after cardiopulmonary bypass
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
ng/mL | 3.08 [1.30 to 6.59] | 3.77 [0.00 to 36.53]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.038, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05

5. Primary Outcome: Plasma Troponin I at 48 Hour After Cardiopulmonary Bypass
Description: Plasma troponin I were measured using enzyme immunoassay (ELISA) in unit of ng/mL
Time Frame: 48 hour after cardiopulmonary bypass
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
ng/mL | 1.66 [0.00 to 7.33] | 1.75 [0.00 to 53.33]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.423, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05

6. Primary Outcome: Plasma Glutamine at Baseline
Description: Plasma glutamine were measured using colorimetric tests in unit of µmol/L
Time Frame: Before induction to anesthesia
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
μmol/L | 555.09 (198.16) | 632.24 (266.36)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.216, Unpaired T-Test — The threshold for statistical significance was p < 0.05

7. Primary Outcome: Plasma Glutamine at 24 Hour After Cardiopulmonary Bypass
Description: Plasma glutamine were measured using colorimetric tests in unit of µmol/L
Time Frame: 24 hour after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
μmol/L | 935.42 (319.10) | 634.79 (243.89)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.001, Unpaired T-Test — The threshold for statistical significance was p < 0.05

8. Secondary Outcome: Right Atrial Appendage Alpha-ketoglutarate
Description: Right atrial appendage alpha-ketoglutarate were measured from right atrial appendage tissue biopsy using colorimetric tests in unit of g/mol.
Time Frame: 5 minute after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: g/mol
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
g/mol | 674.93 (333.49) | 507.32 (280.79)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.043, Unpaired T-Test — The threshold for statistical significance was p < 0.05

9. Secondary Outcome: Right Atrial Appendage Myocardial Injury Score
Description: Right atrial appendage myocardial injury score were measured from tissue section stained with hematoxylin-eosin and examined under by light microscopy in score of 0 (no change) to 3 (major changes with necrosis and diffuse inflammation). Higher scores mean worse outcome
Time Frame: 5 minute after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
score on a scale | 1.30 (0.24) | 1.48 (0.26)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.011, Unpaired T-Test — The threshold for statistical significance was p < 0.05

10. Secondary Outcome: Right Atrial Appendage Apoptosis Index
Description: Right atrial appendage apoptosis index were measured from tissue section stained with in situ terminal deoxynucleotidyl transferase dUTP nick end labelling (TUNEL) and examined under light microscopy in average number of apoptotic cells (positively stained) from 6 random fields per section
Time Frame: 5 minute after cardiopulmonary bypass
Measure: Median (Full Range); unit: cell
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
cell | 5.00 [0.00 to 45.00] | 6.17 [1.00 to 52.00]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.975, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05

11. Secondary Outcome: Anti Cardiac Troponin I Expression
Description: Right atrial appendage anti cardiac troponin I expression were measured from tissue section stained with anti-cardiac troponin I antibody and examined under light microscopy in score of 0 (no change) to -3 (no area observed with anti-cardiac troponin I expression). Higher score mean better outcome
Time Frame: 5 minute after cardiopulmonary bypass
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
score on a scale | -0.33 [-1.00 to 0.00] | -0.83 [-1.00 to 0.00]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p < 0.05

12. Secondary Outcome: Ejection Fraction
Description: Ejection fraction were measured by transesophageal echocardiography using Simpson method in percentage (%)
Time Frame: Immediately after induction of anesthesia
Measure: Median (Full Range); unit: percentage
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
percentage | 41.40 [30.70 to 47.50] | 41.60 [32.00 to 49.60]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.549, Wilcoxon (Mann-Whitney) — The threshold of statistical significance was p < 0.05

13. Secondary Outcome: Ejection Fraction
Description: Ejection fraction were measured by transesophageal echocardiography using Simpson method in percentage (%)
Time Frame: 5 minutes after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
percentage | 46.17 (5.15) | 45.55 (5.03)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.645, Unpaired T-Test — The threshold of statistical significance was p < 0.05

14. Secondary Outcome: Cardiac Index
Description: Cardiac index were measured from pulmonary artery catheter using thermodilution method in unit of L/min/m^2
Time Frame: Immediately after induction of anesthesia, 5 minute, 2 hour, 6 hour, 24 hour after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
L/min/m^2
  Immediately after induction of anesthesia | 2.00 (0.58) | 1.87 (0.35)
  5 minutes after cardiopulmonary bypass | 3.15 (0.57) | 3.03 (0.38)
  2 hours after cardiopulmonary bypass | 2.45 (0.55) | 2.36 (0.56)
  6 hours after cardiopulmonary bypass | 2.54 (0.45) | 2.27 (0.40)
  24 hours after cardiopulmonary bypass | 2.68 (0.35) | 2.47 (0.41)
Statistical Analysis 1: Comparison: Glutamine vs Control; After induction to anesthesia; Test type: Superiority; p = 0.330, Unpaired T-Test — The threshold of statistical significance was p < 0.05
Statistical Analysis 2: Comparison: Glutamine vs Control; 5 minutes after cardiopulmonary bypass; Test type: Superiority; p = 0.352, Unpaired T-Test — The threshold of statistical significance was p < 0.05
Statistical Analysis 3: Comparison: Glutamine vs Control; 2 hours after cardiopulmonary bypass; Test type: Superiority; p = 0.544, Unpaired T-Test — The threshold of statistical significance was p < 0.05
Statistical Analysis 4: Comparison: Glutamine vs Control; 6 hours after cardiopulmonary bypass; Test type: Superiority; p = 0.022, Unpaired T-Test — The threshold of statistical significance was p < 0.05
Statistical Analysis 5: Comparison: Glutamine vs Control; 24 hour after cardiopulmonary bypass; Test type: Superiority; p = 0.038, Unpaired T-Test — The threshold of statistical significance was p < 0.05

15. Secondary Outcome: Plasma Lactate Before Induction to Anesthesia
Description: Plasma lactate were measured using enzymatic method by blood gas analyser machine in unit of mmol/L
Time Frame: Before induction to anesthesia
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
mmol/L | 1.40 [0.90 to 2.40] | 1.30 [0.50 to 2.30]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.200, Wilcoxon (Mann-Whitney) — The threshold of statistical significance was p < 0.05

16. Secondary Outcome: Plasma Lactate 5 Minute After Cardiopulmonary Bypass
Description: Plasma lactate were measured using enzymatic method by blood gas analyser machine in unit of mmol/L
Time Frame: 5 minute after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
mmol/L | 2.02 (0.53) | 2.08 (0.62)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.720, Unpaired T-Test — The threshold of statistical significance was p < 0.05

17. Secondary Outcome: Plasma Lactate 6 Hours After Cardiopulmonary Bypass
Description: Plasma lactate were measured using enzymatic method by blood gas analyser machine in unit of mmol/L
Time Frame: 6 hours after cardiopulmonary bypass
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
mmol/L | 5.30 [1.20 to 9.50] | 5.70 [2.80 to 11.30]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.042, Wilcoxon (Mann-Whitney) — The threshold of statistical significance was p < 0.05

18. Secondary Outcome: Plasma Lactate 24 Hours After Cardiopulmonary Bypass
Description: Plasma lactate were measured using enzymatic method by blood gas analyser machine in unit of mmol/L
Time Frame: 24 hours after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
mmol/L | 2.08 (0.67) | 2.46 (0.69)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.044, Unpaired T-Test — The threshold of statistical significance was p < 0.05

19. Secondary Outcome: Plasma Lactate 48 Hours After Cardiopulmonary Bypass
Description: Plasma lactate were measured using enzymatic method by blood gas analyser machine in unit of mmol/L
Time Frame: 48 hours after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
mmol/L | 2.13 (0.63) | 2.28 (0.61)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.349, Unpaired T-Test — The threshold of statistical significance was p < 0.05

20. Secondary Outcome: Intensive Care Unit Ventilation Time
Description: Intensive care unit ventilation time were measured from length of time participant was on ventilator in intensive care unit in minutes.
Time Frame: 28 days (or until hospital discharge)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
minutes | 652.82 (195.09) | 656.82 (277.07)
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority; p = 0.950, Unpaired T-Test — The threshold of statistical significance was p < 0.05

21. Secondary Outcome: Intensive Care Unit Length of Stay
Description: Intensive care unit length of stay were measured from length of time participant spent in intensive care unit in unit of hours
Time Frame: 28 days (or until hospital discharge)
Measure: Median (Full Range); unit: hours
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
hours | 20.00 [14.00 to 28.00] | 20.00 [16.00 to 29.00]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority — The threshold of statistical significance was p < 0.05; p = 0.862, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Vasoactive Inotropic Score
Description: Vasoactive inotropic score (VIS) were maximum vasoactive and inotropic dose required by participant after surgery measured by VIS=dopamine dose in mg/kgbw/min + dobutamine dose in mg/kgbw/min + 100 x epinephrine dose in mg/kgbw/min + 10 x milrinone dose in mcg/kgbw/min + 10.000 x vasopressin dose in units/kgbw/min + 100 x norepinephrine dose in mcg/kgbw/min. Higher scores means worse outcomes. VIS >= 20 is considered as high VIS and is associated with poor outcomes.
Time Frame: 28 days (or until hospital discharge)
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
score on a scale | 5.00 [0.00 to 15.00] | 5.00 [0.00 to 17.50]
Statistical Analysis 1: Comparison: Glutamine vs Control; Test type: Superiority — The threshold of statistical significance was p < 0.05; p = 0.075, Wilcoxon (Mann-Whitney)

23. Other Pre Specified Outcome: Coronary Graft
Description: Number of coronary arteries grafted during operation
Time Frame: Intraoperative
Measure: Median (Full Range); unit: grafts
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
grafts | 3.00 [2 to 4] | 3.00 [2 to 4]

24. Other Pre Specified Outcome: Total Surgical Procedure Time
Description: Total time taken for the surgical procedure. Measured in minutes.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
minutes | 225.79 (45.60) | 214.48 (50.13)

25. Other Pre Specified Outcome: Cardiopulmonary Bypass Time
Description: Total time measured the patient went under cardiopulmonary bypass. Measured in minutes.
Time Frame: Intraoperative
Measure: Median (Full Range); unit: minutes
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
minutes | 87.00 [55.00 to 113.00] | 78.00 [39.00 to 138.00]

26. Other Pre Specified Outcome: Aortic Cross-clamping Time
Description: Total time the patient underwent aortic cross-clamping during the surgical procedure. Measured in minutes.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glutamine | Control
Number analyzed (Participants) | 29 | 29
minutes | 44.38 (9.07) | 43.86 (14.81)

ADVERSE EVENTS:
Time Frame: 48 hours
Description: No adverse event reported
Arm/Group | Glutamine | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
This study has some limitations. Limitations includes the sampling time of right atrial appendage tissue which was only at 5 minutes after CPB. Right atrial appendage tissue was used for apoptotic index assessment using TUNEL staining. Right atrial appendage tissue could not be sampled at 6 hours after CPB because sternal closure was performed prior to 6 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04560309/Prot_SAP_ICF_000.pdf